CLINICAL TRIAL: NCT06460038
Title: Efficacy and Safety of Tenapanor in Synucleinopathy-Related Constipation
Brief Title: Tenapanor in Synucleinopathy-Related Constipation
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Cedar Valley Digestive Health Center (Other)
Collaborators: Ardelyx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2405-21279
Record Dates: First submitted 2024-06-11; First posted 2024-06-14 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Synucleinopathy; Parkinson's Disease
Keywords: tenapanor; synucleinopathy; Parkinson's disease; constipation
MeSH Terms: conditions — Synucleinopathies; Parkinson Disease; Constipation | interventions — tenapanor

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled trial of tenapanor vs. placebo
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Tenapanor (Experimental): Tenapanor 50 mg orally twice daily for 12 weeks
  Interventions: Drug: Tenapanor
- Placebo (Placebo Comparator): Placebo orally twice daily for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tenapanor — Inhibitor of NHE3
  Arms: Tenapanor
Drug: Placebo — Placebo drug
  Arms: Placebo

SUMMARY:
Investigation of tenapanor as a potential treatment for synucleinopathy-associated constipation

DETAILED DESCRIPTION:
Randomized, double-blind, placebo controlled trial of tenapanor vs. placebo for treating synucleinopathy-associated constipation in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria

1. Age 50-89 years.
2. Diagnosis of PD within Hoehn and Yahr stages 1-3, confirmed by a neurologist per International Parkinson and Movement Disorder Society criteria.
3. Average weekly stool frequency of ≤5 spontaneous bowel movements (SBMs) and ≤2 complete spontaneous bowel movements (CSBMs) over the past 6 months. These criteria will be verified during a 2-week screening period.
4. Stool consistency ≤3 on the Bristol Stool Form Scale (BSFS). This criterion will be verified during a 2-week screening period.
5. Agreement to use contraception, if applicable.

Exclusion Criteria

1. Functional diarrhea or IBS-D/M based on Rome IV Criteria.
2. Symptomatic structural GI abnormalities or inflammatory bowel disease.
3. Significant hepatic (ALT or AST ≥ 2.5x the upper limit of normal) or renal (serum creatinine >2mg/dl) dysfunction.
4. Pregnancy or lactation.
5. Diagnosis of primary dyssynergic defecation by anorectal manometry.

Ages: 50 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Complete spontaneous bowel movements (CSBM) | 6 of 12 weeks
  Our primary endpoint will be CSBM response, defined as an increase of at least one CSBM per week compared to baseline for at least 6 of the 12 treatment weeks. A CSBM is defined as a bowel movement that occurs naturally and is accompanied by a feeling of complete evacuation

SECONDARY OUTCOMES:
Abdominal pain and bloating response | 6 of 12 weeks
  Decrease in severity score of at least 20% or more from baseline in 6 of 12 weeks (pain visual analog scale 1-10 where 10 is worst pain)
Calprotectin | Week 12
  Decrease in fecal calprotectin by 20% or greater
Lipopolysaccharide binding protein | Week 12
  Decrease in serum lipopolysaccharide binding protein by 20% compared to baseline
Complete spontaneous bowel movements (CSBM) continuous | Week 12
  CSBM treated as a continuous variable. The investigators expect an increase of CSBMs in the treatment group compared to the placebo group. A CSBM is defined as a bowel movement that occurs naturally and is accompanied by a feeling of complete evacuation
Plasma zonulin | Week 12
  Decrease in zonulin by 20% compared to baseline

CONTACTS AND LOCATIONS:
Overall Officials: Richard A. Manfready, MD, AM, FACP, Principal Investigator — Cedar Valley Digestive Health Center; Ravindra Mallavarapu, MD, Study Chair — Cedar Valley Digestive Health Center; Harichandana Punukula, PharmD, MS, Study Director — Cedar Valley Digestive Health Center
Locations (1):
- Cedar Valley Digestive Health Center, Waterloo, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified participant data
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Data requests can be submitted starting 6 months after article publication and the data will be made accessible for up to 24 months. Data will be available upon request for 2 years following study publication.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).
URL: https://library.rush.edu/c.php?g=1278924&p=9384947

REFERENCES:
- [Background] Manfready RA, Engen PA, Verhagen Metman L, Sanzo G, Goetz CG, Hall DA, Forsyth CB, Raeisi S, Voigt RM, Keshavarzian A. Attenuated Postprandial GLP-1 Response in Parkinson's Disease. Front Neurosci. 2021 Jul 2;15:660942. doi: 10.3389/fnins.2021.660942. eCollection 2021. PMID 34276285
- [Background] Manfready RA, Forsyth CB, Voigt RM, Hall DA, Goetz CG, Keshavarzian A. Gut-Brain Communication in Parkinson's Disease: Enteroendocrine Regulation by GLP-1. Curr Neurol Neurosci Rep. 2022 Jul;22(7):335-342. doi: 10.1007/s11910-022-01196-5. Epub 2022 May 28. PMID 35633466
- [Background] Post Z, Manfready RA, Keshavarzian A. Overview of the Gut-Brain Axis: From Gut to Brain and Back Again. Semin Neurol. 2023 Aug;43(4):506-517. doi: 10.1055/s-0043-1771464. Epub 2023 Aug 10. PMID 37562457
- [Background] Hall DA, Voigt RM, Cantu-Jungles TM, Hamaker B, Engen PA, Shaikh M, Raeisi S, Green SJ, Naqib A, Forsyth CB, Chen T, Manfready R, Ouyang B, Rasmussen HE, Sedghi S, Goetz CG, Keshavarzian A. An open label, non-randomized study assessing a prebiotic fiber intervention in a small cohort of Parkinson's disease participants. Nat Commun. 2023 Feb 18;14(1):926. doi: 10.1038/s41467-023-36497-x. PMID 36801916
- [Background] Chey WD, Lembo AJ, Rosenbaum DP. Tenapanor Treatment of Patients With Constipation-Predominant Irritable Bowel Syndrome: A Phase 2, Randomized, Placebo-Controlled Efficacy and Safety Trial. Am J Gastroenterol. 2017 May;112(5):763-774. doi: 10.1038/ajg.2017.41. Epub 2017 Feb 28. PMID 28244495
- [Background] Chey WD, Lembo AJ, Yang Y, Rosenbaum DP. Efficacy of Tenapanor in Treating Patients With Irritable Bowel Syndrome With Constipation: A 26-Week, Placebo-Controlled Phase 3 Trial (T3MPO-2). Am J Gastroenterol. 2021 Jun 1;116(6):1294-1303. doi: 10.14309/ajg.0000000000001056. PMID 33337659
- [Background] Chey WD, Lembo AJ, Rosenbaum DP. Efficacy of Tenapanor in Treating Patients With Irritable Bowel Syndrome With Constipation: A 12-Week, Placebo-Controlled Phase 3 Trial (T3MPO-1). Am J Gastroenterol. 2020 Feb;115(2):281-293. doi: 10.14309/ajg.0000000000000516. PMID 31934897